CLINICAL TRIAL: NCT03507725
Title: Improving Patient Experience and Outcomes for Men Undergoing Prostate Biopsy: A Randomized Controlled Trial With Early Stage Consent
Brief Title: Early Staged Consent Before Prostate Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-189
Record Dates: First submitted 2018-04-15; First posted 2018-04-25 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Prostate Cancer
Keywords: mind-body intervention; 18-189
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Meditation; Surveys and Questionnaires

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care + Meditation (Experimental): Usual care (local anaesthesia) + audio-recorded brief mind-dody intervention for 10 minutes before and for 10 minutes during the prostate biopsy procedure
  Interventions: Behavioral: Meditation; Procedure: Prostate Biopsy; Behavioral: Questionnaires
- Usual Care Group (Active Comparator): Time-and-attention control group receiving usual care (local anesthesia) including optional background music in the biopsy procedure room
  Interventions: Procedure: Prostate Biopsy; Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Meditation — The brief mind-body intervention, specifically developed for this study, is a combination of "mindfulness meditation" with a specific cognitive component of "guided imagery". Patient intervention, they will be given headphones connected to an MP4 player in the clinic area to listen to a pre-biopsy mindfulness exercise (10 minutes). They will then be brought into the biopsy procedure room and given a second set of headphones, guiding the patient through the mindfulness intervention during the biopsy procedure (10 minutes).
  Arms: Usual Care + Meditation
Procedure: Prostate Biopsy — Prostate needle biopsy under local anesthesia
Behavioral: Questionnaires — Questionnaires completion will be by telephone interview or manual completion of paper or online REDCap instruments, depending on participant preference.

SUMMARY:
This is a study and a novel approach to clinical trials, testing the feasibility and acceptability of two-stage consent in the context of a trial integrated into routine clinical practice. The investigator will use, as a model, a trial of a brief mind-body intervention) with guided imagery for procedural pain at the time of prostate biopsy. In the two-stage design, patients will first be approached for consent to 1) have their routinely collected clinical data used for research purposes and 2) be randomly selected to be offered an intervention to improve the experience of prostate biopsy. Only patients randomized to the experimental arm will be informed about the benefits and harms of the intervention and will sign a second consent for the experimental treatment. There will be two separate randomizations in this study, one-stage (usual informed consent) vs. two-stage consent and mindfulness intervention vs. control.

ELIGIBILITY:
Inclusion Criteria:

* All male patients that will be scheduled for standard prostate needle biopsy (first, repeat or active surveillance biopsy) under local anesthesia and potentially consented to the mindfulness study of mind-body intervention for prostate biopsy within the next 12 months.
* English fluent

Exclusion Criteria:

* Patient with prior rectal surgery or anal stricture requiring surgical intervention prior to biopsy.
* Prior prostate radiation

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Prostate Cancer
Enrollment: 390 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2024-10-14 (Actual); Study Completion 2024-10-14 (Actual)

PRIMARY OUTCOMES:
number of patients who sign consent form | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Behrar Ehdaie, MD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm